CLINICAL TRIAL: NCT06927362
Title: Effects of Lee Silverman Voice Treatment Big and Dual Task Training on Balance, Cognition and Functional Mobility in Older Adults With Cognitive Impairment.
Brief Title: LSVT Big and Dual Task Training in Cognitive Impaired Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0258 Rabia Aslam
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Impairment; Balance Changes; Cognition Disorders in Old Age; Functional Mobility
Keywords: LSVT big; dual task training; cognitive impaired patients; cognition
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: interventional study model for this study is a parallel-group randomized controlled trial (RCT). This model involves two distinct groups: Group A will receive SLVT BIG intervention and group B will receive cognitive motor dual task training. Warm up and stretching exercises will be done for both groups.
  comparisons between two therapies are unbiased. This parallel structure means each group undergoes its specific intervention throughout the study period without crossover to the other group's intervention. This approach helps assess the difference in effects of the two therapies on balance, cognition and functional mobility in older adults with cognitive impairment.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (LSVT BIG) (Experimental): Group A will receive SLVT BIG intervention for 12 week (4 times per week) for 60 minutes
  Interventions: Other: Lee Silverman treatment big
- Group B ( Dual task training) (Experimental): Group B will receive cognitive motor dual task training for 12 weeks (4 times per week) for 60 minutes.
  Interventions: Other: Dual task training

INTERVENTIONS:
Other: Lee Silverman treatment big — Half of the treatment sessions consist of standardized multidirectional whole-body movements performed with maximal amplitude of reaching and stepping. The second half is designed to address individual deficits in movement that occur in activities of daily living.
  Dosage: 4 consecutive days a week for 12 weeks (16 sessions in one month) for 60 minutes Repetitions: minimum 8-16 repetitions/task
  Arms: Group A (LSVT BIG)
Other: Dual task training — Group B will receive cognitive motor dual task training for 60 minutes, 4 times a week for 12 weeks. The intervention include both motor and cognitive components.
  Arms: Group B ( Dual task training)

SUMMARY:
The goal of this study ifs to determine the comparative effects of Lee Silverman voice treatment Big and dual task training on balance, cognition and functional mobility in older adults with cognitive impairment.

Perform LSVT big four times in a week for about 4 months. Perform dual task training four times in a week for about 4 months. Complete assessments at baseline, the 4th, 8th, 12th weeks, and a follow-up at the 16th week.

Outcome measures include Mini BESTest, MoCA, stroop test and time up and go test. Statistical analyses will assess within-group and between-group effects based on data distribution.

DETAILED DESCRIPTION:
This study, titled "Effects of of lee Silverman voice treatment big and dual task training on balance, cognition and functional mobility in older adults with cognitive impairment" aims to assess the combined effectiveness of Lee Silverman voice treatment and dual task training in older adults with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients.
* Age limit for patients will be above 65.
* Patients with Mild and moderate cognitive impairment patients MoCA 13-25.
* Patients with Berge balance scale value 41-50.
* Patients who give consent to participate in study and undergo relevant test.

Exclusion Criteria:

* Patients with any musculoskeletal disorder in which these exercises are contraindicated.
* Patients using any walking aids.
* Patients with hearing impairment.
* Patients with other neurological conditions with limit the patient participation in planned exercise like stroke, Parkinson's.
* Patients with diagnosed psychiatric disorder or taking medication that affect cognitive function within 24 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Mini BESTest | 4th week
  It is a short form of the BESTest which include 14 items only. The Mini-BESTest includes asses aspects of dynamic balance control also and control while walking and performing a cognitive task.
MoCA (Montreal Cognitive Assessment (For Cognition) | 4th week
  The Montreal Cognitive Assessment (MoCA) is cognitive screening tool which include 30 points. It measures visuospatial, short term memory, orientation, language, executive functioning along with attention/concentration/working memory.
Stroop test | 4th week
  The Stroop task is one of the most widely used measures of cognitive functioning. The Stroop test requires participants to name the color in which a presented word is printed. Numerous studies have shown that participants need more time to name ink colors of incongruent words than to name ink colors of control patches.
Time up and go test | 4th week
  Timed Up and Go (TUG) have been used in clinical settings as a measure of physical performance in older adults with and without cognitive dysfunction. This test requires people to stand up from a chair, walk 3 m, turn around, walk back to the chair, and sit down again.

CONTACTS AND LOCATIONS:
Overall Officials: Arooba Saeed, phD, Principal Investigator — Riphah International University
Locations (1):
- Iqra Medical Complex and Irtiqa Fitness Club, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park MO, Lee SH. Effects of cognitive-motor dual-task training combined with auditory motor synchronization training on cognitive functioning in individuals with chronic stroke: A pilot randomized controlled trial. Medicine (Baltimore). 2018 Jun;97(22):e10910. doi: 10.1097/MD.0000000000010910. PMID 29851819
- [Background] Janssens J, Malfroid K, Nyffeler T, Bohlhalter S, Vanbellingen T. Application of LSVT BIG intervention to address gait, balance, bed mobility, and dexterity in people with Parkinson disease: a case series. Phys Ther. 2014 Jul;94(7):1014-23. doi: 10.2522/ptj.20130232. Epub 2014 Feb 20. PMID 24557655
- [Background] Morris S, Morris ME, Iansek R. Reliability of measurements obtained with the Timed "Up & Go" test in people with Parkinson disease. Phys Ther. 2001 Feb;81(2):810-8. doi: 10.1093/ptj/81.2.810. PMID 11175678
- [Background] Daniel B, Agenagnew L, Workicho A, Abera M. Psychometric Properties of the Montreal Cognitive Assessment (MoCA) to Detect Major Neurocognitive Disorder Among Older People in Ethiopia: A Validation Study. Neuropsychiatr Dis Treat. 2022 Aug 22;18:1789-1798. doi: 10.2147/NDT.S377430. eCollection 2022. PMID 36035074
- [Background] Das S, Mitra K, Mandal M. Sample size calculation: Basic principles. Indian J Anaesth. 2016 Sep;60(9):652-656. doi: 10.4103/0019-5049.190621. PMID 27729692
- [Background] Kim JH, Park JH. Does Cognitive-Physical Dual-Task Training Have Better Clinical Outcomes than Cognitive Single-Task Training Does? A Single-Blind, Randomized Controlled Trial. Healthcare (Basel). 2023 May 25;11(11):1544. doi: 10.3390/healthcare11111544. PMID 37297684
- [Background] Parial LL, Kor PPK, Sumile EF, Leung AYM. Dual-Task Zumba Gold for Improving the Cognition of People With Mild Cognitive Impairment: A Pilot Randomized Controlled Trial. Gerontologist. 2023 Aug 24;63(7):1248-1261. doi: 10.1093/geront/gnac081. PMID 35679826
- [Background] Kaya Aytutuldu G, Ersoz Huseyinsinoglu B, Karagoz Sakalli N, Sen A, Yeldan I. LSVT(R) BIG versus progressive structured mobility training through synchronous telerehabilitation in Parkinson's disease: A randomized controlled trial. Neurol Sci. 2024 Jul;45(7):3163-3172. doi: 10.1007/s10072-024-07322-0. Epub 2024 Jan 25. PMID 38267603
- [Background] Peterka M, Odorfer T, Schwab M, Volkmann J, Zeller D. LSVT-BIG therapy in Parkinson's disease: physiological evidence for proprioceptive recalibration. BMC Neurol. 2020 Jul 11;20(1):276. doi: 10.1186/s12883-020-01858-2. PMID 32652957
- [Background] Huang X, Zhao X, Li B, Cai Y, Zhang S, Wan Q, Yu F. Comparative efficacy of various exercise interventions on cognitive function in patients with mild cognitive impairment or dementia: A systematic review and network meta-analysis. J Sport Health Sci. 2022 Mar;11(2):212-223. doi: 10.1016/j.jshs.2021.05.003. Epub 2021 May 16. PMID 34004389
- [Background] Farhang M, Miranda-Castillo C, Rubio M, Furtado G. Impact of mind-body interventions in older adults with mild cognitive impairment: a systematic review. Int Psychogeriatr. 2019 May;31(5):643-666. doi: 10.1017/S1041610218002302. Epub 2019 Feb 4. PMID 30712518
- [Background] Kim O, Pang Y, Kim JH. The effectiveness of virtual reality for people with mild cognitive impairment or dementia: a meta-analysis. BMC Psychiatry. 2019 Jul 12;19(1):219. doi: 10.1186/s12888-019-2180-x. PMID 31299921
- [Background] Veldkamp R, Baert I, Kalron A, Tacchino A, D'hooge M, Vanzeir E, Van Geel F, Raats J, Goetschalckx M, Brichetto G, Shalmoni N, Hellinckx P, De Weerdt N, De Wilde D, Feys P. Structured Cognitive-Motor Dual Task Training Compared to Single Mobility Training in Persons with Multiple Sclerosis, a Multicenter RCT. J Clin Med. 2019 Dec 10;8(12):2177. doi: 10.3390/jcm8122177. PMID 31835502